CLINICAL TRIAL: NCT05853185
Title: Assessing Success of MTA and Pre-mixed Bioceramic in Mature Teeth With Irreversible Pulpitis With Full Pulpotomy.
Acronym: GCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Sarang Suresh, Principal Investigator, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUMHS/REC/-93
Record Dates: First submitted 2023-03-25; First posted 2023-05-10 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Pulpitis - Irreversible

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pro Root MTA® (Experimental): Patients in this group will receive the pulpotomy with Pro Root MTA®.
  Interventions: Drug: Pro Root MTA®
- EBRRM® (Active Comparator): Patients in this group will receive the pulpotomy with Endosequence Bioceramic Root Repair Material (EBRRM)®.
  Interventions: Drug: EBRRM®

INTERVENTIONS:
Drug: Pro Root MTA® — Patients in this group will receive the pulpotomy with Pro Root MTA®.
  Arms: Pro Root MTA®
Drug: EBRRM® — Patients in this group will receive the pulpotomy with Endo Sequence Bioceramic Root Repair (EBRRM)®.
  Arms: EBRRM®

SUMMARY:
Although many pulpotomy agents are commercially available, there is a dearth of clinical research comparing the efficacy of these agents in treating individuals with irreversible pulpitis. Bioceramic and MTA both have similar clinical uses, but Bioceramic is distinguished from MTA by its superior chemical, physical, and biological properties. This study aims to address this knowledge deficit by assessing the performance of biocompatible materials in pulpotomy procedures for the treatment of symptomatic permanent teeth in adults with deep caries. For permanent teeth with a completed root and a diagnosis of irreversible pulpitis without apical periodontitis, this research will compare the success rates of MTA and EBRRM pulpotomy procedures in order to provide evidence-based clinical practice guidelines for the treatment of this disease.

DETAILED DESCRIPTION:
The goal of this observational study is to test and compare the success of full pulpotomy with Mineral Trioxide Aggregate (MTA) pre-mixed bioceramic in mature teeth with irreversible pulpitis. Participants in this study were patients with irreversible pulpitis without apical periodontal pathosis recruited from the waiting list at the School of Dentistry at Liaquat University of Medical and Health Sciences in Jamshoro. After obtaining informed consent, demographic information, clinical examination results, and binary variables were recorded pre- and intra-operatively. The study's primary aim was to assess postoperative pain, and secondary aims included assessing the presence of swelling, sinusitis, or fistula and detecting tooth mobility. Participants received either MTA or Endo Sequence Bioceramic Root Repair randomly allocated using a lottery system. Follow-up assessments were done initially, after 6 days, and after 6 months, and periapical radiography was done at 6 days and 6 months to detect radiolucency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of irreversible pulpitis without apical periodontitis
2. Either gender
3. Lower Age 10 Years - Upper Age 40 Years

Exclusion Criteria:

* Teeth displaying indications of resorption.
* Teeth that have not fully developed, characterized by open apices.
* Canals that are calcified or obstructed.
* Perforations that were caused by the dentist.
* Fractures in the root
* Teeth that cannot be restored
* • Teeth that are unable to withstand frigid temperatures, have a sinus infection, or have swelling around them.
* There has been no pulp exposure despite the removal of carious lesion.
* Ten minutes after a pulpotomy, hemorrhage could not be stopped.
* Necrotic or partly necrotic pulp is indicated by insufficient bleeding after exposure.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarang Suresh, Principal Investigator — Liaquat University of Medical and Health Science
Locations (1):
- Liaquat University of Medical and Health Sciences, Jāmshoro, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Department of Operative Dentistry & Endodontics, Liaquat University of Medical and Health Sciences, Jamshoro
Pre-assignment Details: All participants fulfilling the inclusion criteria consented for the study.
Period: Overall Study
Arm/Group | Pro Root MTA® | EBRRM®
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall 64 Patients were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pro Root MTA® | EBRRM® | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.19 (10.548) | 31.25 (11.322) | 30.72 (10.868)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 16 | 23 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Clinical Success at 6 Months
Description: Number of participants with clinical success based on following criteria
  * No complaints of pain or discomfort outside of the initial two days following therapy.
  * The tooth shows no signs of pain upon palpation or percussion.
  * A probing pocket depth of less than 4 mm and 1 mm are indicative of normal movement.
  * No inflammation or sinus tract can be seen in the soft tissues around the teeth.
Time Frame: 6 Months
Population: Clinical Outcome Success at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pro Root MTA® | EBRRM®
Number analyzed (Participants) | 32 | 32
Participants | 27 | 30

2. Secondary Outcome: Radiographic Success
Description: Number of participants with clinical success based on absence of Root resorption, furcal pathosis, or fresh periapical pathosis on the radiograph
Time Frame: 6 Months
Population: Patients with no radiographic findings at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pro Root MTA® | EBRRM®
Number analyzed (Participants) | 32 | 32
Participants | 30 | 32

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Pro Root MTA® | EBRRM®
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT05853185/Prot_SAP_ICF_004.pdf